CLINICAL TRIAL: NCT06668298
Title: Clinical Study of G Protein Biased Μ - Opioid Receptor Agonist Oliceridine for Optimizing Postoperative Analgesia Under General Anesthesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HenanPPH-FNN
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Old Age
Keywords: old age; knee arthroplasty; pain
MeSH Terms: conditions — Pain | interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine; Sufentanil

STUDY DESIGN:
Intervention Model Description: All patients who met the inclusion criteria were randomly divided into two groups based on the use of postoperative analgesic pumps: the sufentanil group and the oliceridine group. The sufentanil group received a treatment regimen of sufentanil 2 µ g · kg-1; The treatment regimen for the oliceridine group is oliceridine 0.4mg · kg-1.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oliceridine group (Experimental): Oliceridine 0.4mg · kg-1+tropisetron 10mg, mixed with physiological saline to 100ml. PCIA is set to continuous infusion of 2ml/h, with a single dose of 2ml and a locking time of 15 minutes.
  Interventions: Drug: Oliceridine
- Sufentanil group (Active Comparator): Sufentanil 2 µ g · kg-1+tropisetron 10mg, mixed with physiological saline to 100ml. PCIA is set to continuous infusion of 2ml/h, with a single dose of 2ml and a locking time of 15 minutes.
  Interventions: Drug: Sulfentanil

INTERVENTIONS:
Drug: Oliceridine — The formula for postoperative analgesia pump is oliceridine 0.4mg · kg-1+tropisetron 10mg, mixed with physiological saline to 100ml.
  Arms: Oliceridine group
Drug: Sulfentanil — The analgesic regimen for the sufentanil group is sufentanil 2 µ g · kg-1+tropisetron 10mg, mixed with physiological saline to 100ml.
  Arms: Sufentanil group

SUMMARY:
Traditional opioid analgesia is a treatment method for moderate to severe pain. However, the use of opioid drugs is not without risks. When treating acute pain, patients may experience hypotension, respiratory depression, hypoxia, nausea and vomiting, irritability, and itching. The purpose of this study is to evaluate the comparison of G protein biased μ - opioid receptor agonist oliceridine and traditional μ - opioid receptor agonist sufentanil in terms of analgesia in patients under general anesthesia.

DETAILED DESCRIPTION:
All patients who met the inclusion criteria were randomly divided into two groups based on the use of postoperative analgesic pumps: the sufentanil group and the oliceridine group. The sufentanil group received a treatment regimen of sufentanil 2 µ g · kg-1; The treatment regimen for the oliceridine group is oliceridine 0.4mg · kg-1. The main postoperative observation indicator is the measurement of total pain intensity difference within 48 hours (SPID-48).

ELIGIBILITY:
Inclusion Criteria:

1. Age>65 years old
2. ASA Level I-III
3. BMI 18.5-29.9
4. Patients undergoing knee joint surface replacement surgery under general anesthesia
5. Postoperative Patient Controlled Intravenous Analgesia Pump (PCIA) Treatment
6. Possess reading and writing abilities
7. You can sign an informed consent form

Exclusion Criteria:

1. Suffering from chronic pain or mental illness before surgery
2. Unable to communicate due to cognitive impairment or language barriers before surgery
3. Patients who have used opioid drugs three days before surgery
4. Patients with long-term alcohol consumption
5. Abnormal liver and kidney function or dialysis patients
6. Concurrent severe cardiovascular, respiratory, and autonomic neuropathy
7. Participated in clinical studies of other drugs or medical devices in the past 3 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Measurement of Total Pain Intensity Difference within 48 Hours (SPID-48) | 48hour
  Postoperative pain was evaluated using the NRS Pain Digital Rating Scale at 1, 6, 12, 24, 36, and 48 hours post surgery; Multiply the difference in pain intensity at each post baseline time point within 48 hours (subtracting the pain intensity at a specific post baseline time point from the pain intensity at baseline) by the duration (in hours) of the previous time point, and then add them up.

SECONDARY OUTCOMES:
Adverse reactions | 48hour
  Incidence of nausea, vomiting, dizziness, headache, constipation, itching, and hypoxia

CONTACTS AND LOCATIONS:
Overall Officials: Jiaqiang Zhang, Study Director — Chief physician

IPD SHARING:
Plan to Share IPD: No